CLINICAL TRIAL: NCT04576611
Title: Behavioral Activation and Exercise Protocol for Chronic Pain Patients Based on the Use of New Technologies (Smartphone)
Brief Title: LOw Level of Activity (LOLA): Education and Exercise-based Intervention for Low Back Pain
Acronym: LOLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSI2015-66295
Record Dates: First submitted 2020-07-10; First posted 2020-10-06 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Low Back Pain
Keywords: Mobile Applications; Muscle and Stretching Exercises; Physical Exercise; Behavior
MeSH Terms: conditions — Low Back Pain; Motor Activity; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- face-to-face (Experimental): A 4-week intervention (8 sessions) will be carried out in a group of patients with non-specific chronic low back pain using face-to-face modality guided by a health professional.
  Interventions: Other: face-to-face protocol
- self-managed (Experimental): A 4-week intervention (8 sessions) will be carried out in a group of patients with non-specific chronic low back pain using self-managed modality through BackFit App.
  Interventions: Other: self-managed protocol

INTERVENTIONS:
Other: face-to-face protocol — The intervention is based on education (on pain neurophysiology and healthy lifestyle habits) and physical exercise (strength, flexibility, joint mobility and self-massage).
  Arms: face-to-face
Other: self-managed protocol — Subjects of this group receive the same intervention content as the other experimental group, but through a mobile application.
  Arms: self-managed

SUMMARY:
Chronic pain of moderate to severe intensity occurs in 19% of adult Europeans. Non-specific low-back pain is one of the most prevalent symptoms and the main cause of disability in industrialized countries, generating significant public health expenditure on health and occupational care. The combination of pain neurophysiology education and therapeutic exercise has shown positive effects in patients with chronic non-specific low back pain. Mobile health tools (mHealth) are proposed as a cost-effective alternative to continuously record the daily activities of patients and to provide rapid feedback to users and clinicians, reducing visits to clinics. A 4-week (8-session) education and exercise-based intervention will be carried out in a group of patients with non-specific chronic low back pain using two modalities: (1) face-to-face guided by a health professional or (2) self-managed through BackFit App. The sample will be divided into two groups and will be evaluated before (pre), after (post) and 3 months (follow-up) after the intervention.

DETAILED DESCRIPTION:
The objectives of this study are:

1. To assess the influence of a 4-week (8 sessions) intervention based on education (about pain neurophysiology and healthy lifestyle habits) and physical exercise (strength, flexibility, joint mobility, and self-massage) on pressure pain thresholds (PPT) and cognitive functioning (selective attention), as primary variable outcomes, and on physical condition (balance and range of movement), affective and cognitive symptoms (mood, anxiety, catastrophizing, fear-avoidance beliefs and kinesiophobia), pain interference and self-reported clinical pain, as secondary variable outcomes, in patients with non-specific chronic low back pain.
2. To evaluate the effectiveness of a mobile health application developed by researchers (BackFit App) to carry out the intervention, in comparison with a supervised intervention by a health professional.

The hypotheses of the study are:

1. This intervention based on education and physical exercise will increase PPT and improve selective attention.
2. This intervention will also improve physical condition, self-reported clinical pain, affective and cognitive symptoms and pain interference presented by patients with chronic low back pain.
3. The intervention performed with BackFit App will be as effective as that supervised by a health professional.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 18 and 59 years, with non-specific low back pain for more than 6 weeks and which have experienced at least 3 episodes of low back pain lasting more than 1 week during the year prior to the study, and, at the time of evaluation and/or intervention, presenting pain of mild/moderate intensity (not exceeding 5 out of 10 in a Visual Analogue Scale (VAS)).

Exclusion Criteria:

* High functional impairment compromising activities such as walking, sitting or getting up from a chair.
* Pain at the time of evaluation and/or intervention greater than 5 (out of 10) in a VAS.
* Presence of irradiated pain (sciatic type) or referred to lower extremities.
* History of spine surgery, spinal or pelvic fracture
* Hospitalization for serious trauma or injuries due to traffic accidents.
* History of osteoarthritis in the lower extremities.
* History of any systematic diseases with involvement of the locomotor system.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 59 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Cognitive functioning assessment. | Up to 4 weeks.
  Cognitive functioning was assessed by recording electroencephalographic activity during a computerized version of the Flanker task, which measures selective attention, under two experimental conditions: congruent flanks (arrows) with the target (pointing in the same direction as the central arrow) and incongruent (pointing the opposite direction).Regarding Resting EEG a Fast Fourier Transform (FFT) analysis has been made (delta, theta, "Alpha" and beta 1, 2 and 3. The EEG during the "Flanker task" was analyzed by means of a "Cluster-based analysis". Primary outcome measures were recorded in a counterbalanced order and were measured at baseline and 4 weeks.
Heart Rate Variability (HRV) | Up to 4 weeks.
  Heart Rate Variability (HRV) has been analyzed from ECG data. Primary outcome Measures were recorded in a counterbalanced order and were measured at baseline and 4 weeks.
Pressure pain thresholds (PPT). | Up to 12 weeks.
  To evaluate Pressure pain thresholds (PPT )(with a maximum of 5kg/cm2) will be applied pressure on the erector spinae and index finger with an algometer (area 1cm2). Primary outcome measures were recorded in a counterbalanced order and were measured at baseline, 4 and 12 weeks.

SECONDARY OUTCOMES:
Balance | Up to 12 weeks.
  Mono and bipedal static balance will be measured with the Wii balance board. Measurements will be performed after 15 minutes of rest once the subject arrives at baseline, 4 and 12 weeks.
Range of movement | Up to 12 weeks.
  Range of movement of the hip will be measured with a goniometer. Measurements will be performed after balance measurements at baseline, 4 and Range of movement of the hip will be measured with a goniometer. Measurements will be performed after balance measurements at baseline, 4 and 12 weeks.
Clinical pain | Up to 12 weeks.
  Clinical pain will be measured with Visual Analog Scale (VAS) (0-10cm) This outcome was measured at baseline, 4 and 12 weeks. A higher score indicates greater pain intensity.
Pain interference | Up to 12 weeks.
  Pain interference data will be collected with the Spanish version of Oswestry Disability Index (ODI) (0-100%). This outcome was measured at baseline, 4 and 12 weeks. A higher score indicates greater functional disability.
Affective symptoms (Mood) | Questionnaires will be performed during rest prior to balance and range of movement measurements at baseline, 4 and 12 weeks
  Mood, often associated to chronic pain, will be assessed by the Spanish versions of Profile of Mood States (POMS) questionnaire.
  The POMS questionnaire (Ranges from 0-200) assesses six mood subscales: tension-anxiety (0-36), anger-hostility (0-48), vigor (0-32), fatigue (0-28), depression (0-60) and confusion (0-28).
  High vigor scores reflect a good mood or emotion. Low scores in the other subscales reflect a good mood or emotion
Affective symptoms (anxiety) | Questionnaires will be performed during rest prior to balance and range of movement measurements at baseline, 4 and 12 weeks
  Anxiety, often associated to chronic pain, will be assessed by the State Trait Anxiety Inventory (STAI) questionnaire. State (0-30) and Trate (0-30). Higher scores indicates greater anxiety.
Cognitive symptoms (catastrophizing) | Questionnaires will be performed during rest prior to balance and range of movement measurements at baseline, 4 and 12 weeks
  Other cognitive symptoms, such as catastrophyzing, will be assessed using the Spanish version of Pain Catastrophizing Scale (PCS)(Ranges from 0-52), a 13-item scale where low scores show little catastrophization, and high values, high catastrophization.
Cognitive symptoms (fear-avoidance beliefs) | Questionnaires will be performed during rest prior to balance and range of movement measurements at baseline, 4 and 12 weeks
  Other cognitive symptoms, such as fear-avoidance beliefs will be also assessed using Fear Avoidance Beliefs Questionnaire (FABQ).(ranges from 0-96) Higher scores indicate more strongly held fear avoidance beliefs.
Cognitive symptoms (kinesiophobia) | Questionnaires will be performed during rest prior to balance and range of movement measurements at baseline, 4 and 12 weeks
  Other cognitive symptoms, such as kinesiophobia (or fear of movement) will be also assessed using the spanish version of Tampa Scale for Kinesiophobia (TSK).
  It consists of 11 items scored from 1 (strongly disagree) to 4 (strongly agree). The higher the score, the higher the degree of kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Sitges, PhD, Principal Investigator — University of Balearic Islands, Department of Psychology
Locations (1):
- University of the Balearic Islands, Palma, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Breivik H, Collett B, Ventafridda V, Cohen R, Gallacher D. Survey of chronic pain in Europe: prevalence, impact on daily life, and treatment. Eur J Pain. 2006 May;10(4):287-333. doi: 10.1016/j.ejpain.2005.06.009. Epub 2005 Aug 10. PMID 16095934
- [Background] van Tulder M, Becker A, Bekkering T, Breen A, del Real MT, Hutchinson A, Koes B, Laerum E, Malmivaara A; COST B13 Working Group on Guidelines for the Management of Acute Low Back Pain in Primary Care. Chapter 3. European guidelines for the management of acute nonspecific low back pain in primary care. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S169-91. doi: 10.1007/s00586-006-1071-2. No abstract available. PMID 16550447
- [Background] Delitto A, George SZ, Van Dillen L, Whitman JM, Sowa G, Shekelle P, Denninger TR, Godges JJ; Orthopaedic Section of the American Physical Therapy Association. Low back pain. J Orthop Sports Phys Ther. 2012 Apr;42(4):A1-57. doi: 10.2519/jospt.2012.42.4.A1. Epub 2012 Mar 30. PMID 22466247
- [Background] Bardin LD, King P, Maher CG. Diagnostic triage for low back pain: a practical approach for primary care. Med J Aust. 2017 Apr 3;206(6):268-273. doi: 10.5694/mja16.00828. PMID 28359011
- [Background] Bodes Pardo G, Lluch Girbes E, Roussel NA, Gallego Izquierdo T, Jimenez Penick V, Pecos Martin D. Pain Neurophysiology Education and Therapeutic Exercise for Patients With Chronic Low Back Pain: A Single-Blind Randomized Controlled Trial. Arch Phys Med Rehabil. 2018 Feb;99(2):338-347. doi: 10.1016/j.apmr.2017.10.016. Epub 2017 Nov 11. PMID 29138049
- [Background] Nijs J, Lluch Girbes E, Lundberg M, Malfliet A, Sterling M. Exercise therapy for chronic musculoskeletal pain: Innovation by altering pain memories. Man Ther. 2015 Feb;20(1):216-20. doi: 10.1016/j.math.2014.07.004. Epub 2014 Jul 18. PMID 25090974
- [Background] Dobkin BH, Dorsch A. The promise of mHealth: daily activity monitoring and outcome assessments by wearable sensors. Neurorehabil Neural Repair. 2011 Nov-Dec;25(9):788-98. doi: 10.1177/1545968311425908. PMID 21989632
- [Derived] Sitges C, Terrasa JL, Garcia-Dopico N, Segur-Ferrer J, Velasco-Roldan O, Crespi-Palmer J, Gonzalez-Roldan AM, Montoya P. An Educational and Exercise Mobile Phone-Based Intervention to Elicit Electrophysiological Changes and to Improve Psychological Functioning in Adults With Nonspecific Chronic Low Back Pain (BackFit App): Nonrandomized Clinical Trial. JMIR Mhealth Uhealth. 2022 Mar 15;10(3):e29171. doi: 10.2196/29171. PMID 35289758